CLINICAL TRIAL: NCT02615535
Title: Neurofeedback-enhanced Mindfulness Meditation for the Treatment of Affective and Attentional Disturbances in Patients With Traumatic Brain Injury
Brief Title: Neurofeedback-enhanced Mindfulness Meditation in Traumatic Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spaulding Rehabilitation Hospital (Other)
Collaborators: InteraXon, Inc. (Industry)
Responsible Party: Principal Investigator, Mel B. Glenn, Director of Outpatient and Community Brain Injury Rehabilitation, Spaulding Rehabilitation Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015P002184
Record Dates: First submitted 2015-11-18; First posted 2015-11-26 (Estimated); Results first posted 2019-12-06 (Actual); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Traumatic Brain Injury
Keywords: traumatic brain injury
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Neurofeedback

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- EEG neurofeedback-assisted meditation (Experimental): EEG neurofeedback assisted meditation using the MUSE device and auditory feedback.
  Interventions: Device: EEG neurofeedback-assisted meditation
- Non-EEG feedback-assisted meditation (Active Comparator): Non-EEG neurofeedback assisted meditation. Subjects will have auditory instruction from the MUSE device without the EEG neurofeedback.
  Interventions: Device: Non-EEG feedback-assisted meditation

INTERVENTIONS:
Device: EEG neurofeedback-assisted meditation — meditation with auditory feedback regarding EEG status
  Other Names: MUSE
  Arms: EEG neurofeedback-assisted meditation
Device: Non-EEG feedback-assisted meditation — meditation without auditory feedback regarding EEG status
  Other Names: MUSE without EEG feedback
  Arms: Non-EEG feedback-assisted meditation

SUMMARY:
Spaulding Rehabilitation Hospital is conducting a research study evaluating the effectiveness of the brain-training product, MUSE, an EEG-guided neurofeedback device designed to assist in cultivating a relaxed, attentive state of mind during meditation. The investigators study aims to evaluate whether such a tool could be useful in treating persistent traumatic brain injury symptoms such as inattention, impulsivity, irritability, or dysregulated mood.

DETAILED DESCRIPTION:
Twenty subjects in total will participate in this study. Subjects will be randomized to focused-attention meditation training with or without the neurofeedback device, MUSE. Subjects will be asked to practice ~10 min of daily meditation for 6-8 weeks. Neuropsychological testing will be performed at the beginning of the study and after six weeks of training. At this time point, those randomized to the non-MUSE group will be given a device and asked to train for an additional two weeks. At the conclusion of the study, all subjects will also undergo a brief telephone or in-person exit interview regarding their experiences using the MUSE device.

Primary endpoint: change in Neurobehavioral Symptom Inventory

Secondary endpoints: change in the following: Wechsler Adult Intelligence Scale-IV Digit Span and Symbol-Digit Coding, Trail-Making Test, Beck Anxiety Inventory, Beck Depression Inventory, Cognitive and Affective Mindfulness Scale-Revised, percentage of EEG activity associated with alpha, beta, or theta activity.

ELIGIBILITY:
Inclusion Criteria:

1. history of mild-moderate traumatic brain injury
2. impaired attention or concentration
3. >1 year since traumatic brain injury
4. ability to participate in neurofeedback and mindfulness meditation
5. daily access to a smart phone
6. on stable dosage of neuropsychological medications with no significant changes planned for the duration of the study
7. no prior history of a meditation practice

Exclusion Criteria:

1. severe mental illness or psychological symptoms (severe depression, suicidality, disabling anxiety, PTSD, psychosis, dissociation)
2. significant pre-morbid learning disability
3. current or recent (in past year) history of significant drug or alcohol abuse
4. medical illness severe enough to result in an attentional disorder
5. neurodegenerative disease
6. non-fluency in English.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2019-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mel B Glenn, MD, Principal Investigator — Spaulding Rehabilitation Hospital
Locations (1):
- Spaulding Rehabilitation Hospital Boston, Charlestown, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
If participants request their outcome data, we will provide this to them with a brief discussion of its meaning and limitations on interpretation.

REFERENCES:
- [Background] Brandmeyer T, Delorme A. Meditation and neurofeedback. Front Psychol. 2013 Oct 7;4:688. doi: 10.3389/fpsyg.2013.00688. eCollection 2013. No abstract available. PMID 24109463
- [Background] Chiesa A, Calati R, Serretti A. Does mindfulness training improve cognitive abilities? A systematic review of neuropsychological findings. Clin Psychol Rev. 2011 Apr;31(3):449-64. doi: 10.1016/j.cpr.2010.11.003. Epub 2010 Dec 1. PMID 21183265
- [Background] Cicerone KD, Langenbahn DM, Braden C, Malec JF, Kalmar K, Fraas M, Felicetti T, Laatsch L, Harley JP, Bergquist T, Azulay J, Cantor J, Ashman T. Evidence-based cognitive rehabilitation: updated review of the literature from 2003 through 2008. Arch Phys Med Rehabil. 2011 Apr;92(4):519-30. doi: 10.1016/j.apmr.2010.11.015. PMID 21440699
- [Background] Hofmann SG, Sawyer AT, Witt AA, Oh D. The effect of mindfulness-based therapy on anxiety and depression: A meta-analytic review. J Consult Clin Psychol. 2010 Apr;78(2):169-83. doi: 10.1037/a0018555. PMID 20350028
- [Derived] Polich G, Gray S, Tran D, Morales-Quezada L, Glenn M. Comparing focused attention meditation to meditation with mobile neurofeedback for persistent symptoms after mild-moderate traumatic brain injury: a pilot study. Brain Inj. 2020 Aug 23;34(10):1408-1415. doi: 10.1080/02699052.2020.1802781. Epub 2020 Aug 12. PMID 32783645

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | EEG Neurofeedback-assisted Meditation | Non-EEG Feedback-assisted Meditation
Started | 14 | 11
Completed | 10 | 10
Not Completed | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | EEG Neurofeedback-assisted Meditation | Non-EEG Feedback-assisted Meditation | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 20
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.3 (3.6) | 41.4 (4.7) | 45.4 (3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 17
  Male | 1 | 2 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 10 | 9 | 19
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Change in Neurobehavioral Symptom Inventory
Description: Measures common symptoms after head injury. This scales ranges from 0-4 on 22 items, for a minimum score of 0 and a maximum score of 88. Higher scores mean a greater severity of symptoms.
Time Frame: baseline and six weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | EEG Neurofeedback-assisted Meditation | Non-EEG Feedback-assisted Meditation
Number analyzed (Participants) | 10 | 10
units on a scale
  baseline | 35.2 (3) | 33.1 (5.1)
  6 weeks | 27.7 (2.8) | 24.6 (3.9)

2. Secondary Outcome: Change in Wechsler Adult Intelligence Scale-IV Digit Span
Description: Tests participants digit span, repeating forward sequences of digits from 2 to 8. Scale ranges from 0 to 16. Higher scores mean a better outcome.
Time Frame: baseline and six weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | EEG Neurofeedback-assisted Meditation | Non-EEG Feedback-assisted Meditation
Number analyzed (Participants) | 10 | 10
units on a scale
  baseline | 10.4 (0.7) | 11.2 (1)
  six weeks | 10.9 (0.6) | 11.8 (0.8)

3. Secondary Outcome: Change in Wechsler Adult Intelligence Scale-IV Digit Symbol Coding
Description: A subject is provided with a key matching nine numbers to nine unique symbols. Numbers are then provided in random order and subjects have 120 seconds to match as many numbers with symbols as possible. All correct responses are scored. Scores range from 0 to 135. Scores are later scaled from 1 to 19. Higher scores mean a better outcome.
Time Frame: baseline and six weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | EEG Neurofeedback-assisted Meditation | Non-EEG Feedback-assisted Meditation
Number analyzed (Participants) | 10 | 10
units on a scale
  baseline | 11.6 (1.2) | 11.1 (0.9)
  six weeks | 13.1 (1.1) | 12.5 (0.8)

4. Secondary Outcome: Change in Trail Making Test
Description: Subjects are asked to sequence numbers and letters represented on a page as quickly as then can. Results are measured in seconds, ranging from 0 (hypothetically) to an infinite number (hypothetically). Results are scaled from 1 to 19. Lower scores mean a better outcome.
Time Frame: baseline and six weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | EEG Neurofeedback-assisted Meditation | Non-EEG Feedback-assisted Meditation
Number analyzed (Participants) | 10 | 10
units on a scale
  baseline | 10.9 (1) | 11.9 (0.4)
  six weeks | 12.3 (0.8) | 12.7 (0.4)

5. Secondary Outcome: Change in Beck Anxiety Inventory
Description: Subjects rate on a 0-3 likert scales responses to questions about anxiety. Scores range from 0-63. Lower scores mean a better outcome.
Time Frame: baseline and six weeks
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | EEG Neurofeedback-assisted Meditation | Non-EEG Feedback-assisted Meditation
Number analyzed (Participants) | 10 | 10
score on a scale
  baseline | 15.9 (1.9) | 18.8 (4.6)
  six weeks | 11.5 (1.9) | 8.5 (1.8)

6. Secondary Outcome: Change in Beck Depression Inventory-II
Description: Subjects respond to questions on a Likert scale from 0-3 regarding depressive symptoms. There are 21 items. Scores range from 0-63. Lower scores mean a better outcome.
Time Frame: baseline and six weeks
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | EEG Neurofeedback-assisted Meditation | Non-EEG Feedback-assisted Meditation
Number analyzed (Participants) | 10 | 10
score on a scale
  baseline | 19.9 (3.6) | 17 (3.5)
  six weeks | 13.1 (3.1) | 9.9 (2.8)

7. Secondary Outcome: Change in Cognitive and Affective Mindfulness Scale-Revised
Description: Subjects answer questions regarding mindfulness on a Likert Scale from 1-4. There are twelve questions total. Scores range from 4-48. Higher scores mean a better outcome.
Time Frame: baseline and six weeks
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | EEG Neurofeedback-assisted Meditation | Non-EEG Feedback-assisted Meditation
Number analyzed (Participants) | 10 | 10
score on a scale
  baseline | 24.2 (2) | 24.7 (1.8)
  six weeks | 27.3 (1.6) | 28.3 (2.1)

8. Secondary Outcome: Change in Percentage of EEG Activity Associated With Alpha, Beta, and Theta Rhythms as Measured by Surface Electrodes on the MUSE Device
Description: Change in "percent Calm" as determined by Muse device. Equations behind this algorithm to determine "Calm" are proprietary and were not shared by the device manufacturer. Ranges from 0% to 100%. Higher scores mean a better outcome.
Time Frame: baseline and at six weeks
Measure: Mean (Standard Error); unit: percentage of "Calm"
Arm/Group | EEG Neurofeedback-assisted Meditation | Non-EEG Feedback-assisted Meditation
Number analyzed (Participants) | 10 | 10
percentage of "Calm"
  baseline | 49.7 (5.6) | 32 (7.8)
  six weeks | 57.7 (7.6) | 43.7 (9.9)

ADVERSE EVENTS:
Time Frame: Adverse effects from meditation were not anticipated. Subjects practiced meditation for six weeks each. If adverse effects occurred during the six weeks, they contacted our group. At our post-intervention assessment at six weeks, we asked specifically about adverse events. Adverse events were not monitored beyond the intervention period of six weeks.
Description: Definitions are consistent.
Arm/Group | EEG Neurofeedback-assisted Meditation | Non-EEG Feedback-assisted Meditation
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-01): https://cdn.clinicaltrials.gov/large-docs/35/NCT02615535/Prot_SAP_000.pdf